CLINICAL TRIAL: NCT04451590
Title: Virtual Reality: a Teaching-learning Strategy for Cognitive Mastery in Airway Trauma
Brief Title: Virtual Reality: a Teaching-learning Strategy for Cognitive Mastery in Airway Trauma Management
Acronym: AW&VR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 108-2019
Record Dates: First submitted 2019-11-12; First posted 2020-06-30 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Education, Medical; Airway Management; Students, Medical; Virtual Reality; Trauma Centers; Manikins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An external assessor will score videos participants performing Airway Trauma Management using the Airway Injury Checklist on Core Decision Making Steps. The assessors will be blinded to intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-based Simulation (Intervention) (Experimental): Students will receive training on traumatic airway management using VR-based simulation.
  Interventions: Other: VR-based simulation
- Mannequin-based Simulation (Control) (Other): Students will receive training on traumatic airway management using mannequin-based simulation.
  Interventions: Other: Mannequin-based simulation

INTERVENTIONS:
Other: VR-based simulation — Participants will experience a novel interactive and immersive VR full size trauma bay with an adult patient and healthcare professionals. Immersed in the environment, learners undertake the decision-making steps in managing the medical care for a patient with an airway injury. Learners are first given the case scenario from which they form their own learning goals/plans. They then navigate through the scenario that will provide feedback depending on their actions in the form of either the patient's hemodynamic changes or prompts from healthcare avatars in the scenario. These feedback processes are built-in and designed to promote reflection and reorganization of the learner's decision-making strategies. As learning progresses, fewer prompts will be given. At the end of the scenario, evaluation algorithms pre-programmed into the VR-based simulation will be displayed.
  Arms: VR-based Simulation (Intervention)
Other: Mannequin-based simulation — Participants will experience a mannequin-based scenario practice which is the current gold standard in medical education. The trauma airway management scenario will match the VR environment and sequence of events.
  Arms: Mannequin-based Simulation (Control)

SUMMARY:
Airway injury in patients is a high risk and complex medical crisis. Unfortunately, training for airway management in injured patients is challenging. The most effective way of practicing airway management is using mannequins. However, mannequin training is expensive and only occasionally available to medical trainees.

The purpose of this study is to determine if Virtual Reality (VR) can be used to educate medical students on airway injury management. VR training will involve managing the care of a patient with an airway injury in an immersive, interactive VR hospital trauma bay. The investigators will compare the knowledge gained from VR training vs. mannequin training. The investigators will also investigate whether VR training teaches students faster than mannequin training. In addition, the investigators will identify factors which might affect learning from VR.

Medical students who choose to participate will be randomized (i.e. participant will have a 50% chance to be placed in either group) to be trained with VR or a mannequin. Participants then will be trained on airway injury management using their assigned training approach. One week later, all participants will be assessed on their airway injury management skills using a mannequin. Before and after their sessions, participants will also be asked to complete a questionnaire on their clinical decision-making. Participants who received VR training will also complete a questionnaire about their experience with the VR training.

This study will help develop a new approach to airway management training which is cheaper and more easily available to medical trainees than mannequin training. This educational tool could lead to better treatment of airway trauma in future patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 at time of consent
* Medical student at U of T in 1st, 2nd or 3rd year
* Able to attend two sessions a week apart

Exclusion Criteria:

* Lack of participant consent or capacity to give consent
* History of significant motion sickness (during exposure to physical, visual and virtual motion, cybersickness verbally declared by patient)
* Visual/hearing impairments that affect abilities to listen/watch videos/VR video

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Traumatic Airway Injury Management Knowledge | up to 24 hours before and up to 24 hours after practice sessions
  Knowledge acquisition of traumatic airway injury management as assessed by the written Key Features Decision Making Checklist, Change from baseline (pre-training) knowledge to after practice session knowledge (post-training).
Application of Traumatic Airway Injury Management Knowledge | 7 days after practice session
  Application of decision making concepts surrounding traumatic airway injury management as assessed by the Airway Injury Checklist of Core Decision Making Steps completed during participant performance of a simulated crisis assessment scenario.

SECONDARY OUTCOMES:
Number of Required Practice Sessions | During the 1 day practice session
  Identify whether VR or mannequin-based simulation practice require fewer practice sessions to achieve learning objectives.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data will be made available upon reasonable request to study PI following publication of full trial results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available following publication.
Access Criteria: Data and supporting information will be made available following reasonable request directly to study PI.